CLINICAL TRIAL: NCT02224911
Title: Use of Laser Interstitial Thermal Therapy in the Focal Treatment of Localized Prostate Cancer: A Pilot Feasibility Study
Brief Title: Use of Laser Interstitial Thermal Therapy in the Focal Treatment of Localized Prostate Cancer
Acronym: LITT
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-000409; JCCCID436 (Other: Jonsson Comprehensive Cancer Center); NCI-2015-01487 (Other: CTRP)
Record Dates: First submitted 2014-07-21; First posted 2014-08-25 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: focal therapy; prostate cancer treatment; laser treatment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Laser Interstitial Thermal Therapy: This is a minimally invasive procedure for focal treatment of prostate cancer.
  Interventions: Device: Laser Interstitial Thermal Therapy

INTERVENTIONS:
Device: Laser Interstitial Thermal Therapy

SUMMARY:
This is a pilot, feasibility/exploratory study to evaluate the safety of laser interstitial thermal therapy (LITT) using Visualase in the focal treatment of localized prostate cancer as well as to gather data for the design of future studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with initial presentation of organ confined prostate cancer (clinical stage ≤ T2b)

  * Negative metastatic workup with bone scan and CT abdomen/pelvis, within 6 months of study treatment, if indicated by PSA >10
  * Age 40 years to 85 years of age
  * Multi-parametric MRI at UCLA within 6 months of study treatment, demonstrating a

    * Region of interest (ROI) of MRI suspicion level 3 or higher
    * ROI located proximal to the external sphincter by a margin of at least 2 cm
  * Transrectal ultrasound-guided biopsy with ≥ 10 systematic biopsy cores and ≥ 2 MRI-ultrasound fusion targeted biopsy cores from above MRI-derived ROI

    * Histologically-confirmed adenocarcinoma from targeted biopsy cores (≥ 2 cores)
    * Overall Gleason score not to exceed 3+4
  * Subjects desire focal therapy and declined conventional treatment (active surveillance, radical prostatectomy, radiation therapy, cryosurgery and hormone therapy)
  * Signed informed consent for the LITT treatment through the 12 month follow up visit

Exclusion Criteria:

* Any significant cancer outside of MRI target (ROI) area, defined as Gleason score > 3+4
* < 10 years life expectancy
* American Society of Anesthesiologists (ASA) criteria of IV or higher
* Unfit for conscious sedation anesthesia
* Active bleeding disorder as determined by abnormal prothrombin time, partial thromboplastin time, INR or platelet count (as determined by institutional lab parameters) at the time of screening
* Use of coumadin or any other anticoagulant, unless anticoagulation can be temporarily reversed or stopped for a window of at least 7 days peri-procedure
* Active urinary tract infection
* Prostate abscess, chronic or acute prostatitis, or neurogenic bladder
* Any prior treatment for prostate cancer

  * Radical prostatectomy
  * Radiation therapy (external beam or brachytherapy)
  * Cryotherapy
  * High intensity focused ultrasound treatment
  * Photodynamic therapy
  * Androgen deprivation therapy
* Prior prostate, bladder neck, or urethral stricture surgery

  * Any prostate debulking procedure, including: transurethral resection of prostate, photovaporization, or electrovaporization
  * Transurethral incision of bladder neck
  * Urethral stricture dilation or reconstruction
* Any current 5-alpha reductase inhibitors (history of use ≥ 6 months prior to MRI is acceptable)
* Prior significant rectal surgery (hemorrhoidectomy is acceptable)
* Rectal fissure, fibrosis, stenosis, or other anatomic abnormality precluding insertion of transrectal device
* History of inflammatory bowel disease
* Urinary tract or rectal fistula
* Any contraindication to MRI (contrast allergy severe claustrophobia, MRI-incompatible prosthesis)

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men, 40 to 85 years of age, recently diagnosed with prostate cancer using the MRI fusion technology.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 12 months

SECONDARY OUTCOMES:
Absence of prostate cancer in the MRI target area as measure of efficacy. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pantuck Alan, MD, Principal Investigator — University of California, Los Angeles; Steven Raman, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Carter HB, Kettermann A, Warlick C, Metter EJ, Landis P, Walsh PC, Epstein JI. Expectant management of prostate cancer with curative intent: an update of the Johns Hopkins experience. J Urol. 2007 Dec;178(6):2359-64; discussion 2364-5. doi: 10.1016/j.juro.2007.08.039. Epub 2007 Oct 22. PMID 17936806